CLINICAL TRIAL: NCT06390085
Title: Optical Measurements of the Skin Surface to Infer Distinctions in Myofascial Tissue Stiffness
Acronym: OptMeasSkin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gregory J. Gerling, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRBSBS6201; 5U24AT011969 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-04-30 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Tissue Pain
Keywords: myofascial tissue; skin surface; optical imaging; deformation
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Intervention Model Description: Evaluating objective imaging biomarkers for characterizing myofascial pain and mobility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual therapy intervention (Experimental): Those participants with myofascial pain in the cervicothoracic region are assessed by manual palpation by a trained clinician.
  Interventions: Other: Soft tissue manipulation

INTERVENTIONS:
Other: Soft tissue manipulation — The clinician will perform a soft tissue massage intervention where she/he will use moderate massaging and compression. The amount of pressure is less than 5 N, the velocity is low at a controlled rate of 1 Hz, the duration of 30 seconds, angle 90 and 45 degrees.

SUMMARY:
This study involves imaging the skin movements of surface tissue on the back. A clinician will perform assessment and intervention procedures manually, using manual and light movements of stretch and compression.

DETAILED DESCRIPTION:
This study includes a demographic questionnaire, self-report on level of pain, application of ink to the skin, manual clinical assessments, and a massage intervention. The study will take place entirely in Olsson Hall. All information collected will be recorded using a randomized identification number.

1. Upon arrival for the study, a participant will be asked to read, review, and sign this informed consent agreement.
2. Next, the participant will be asked verbally to complete a demographic questionnaire.
3. The study team will verbally ask the participant to rate the current level of pain.
4. The participant will have been asked to bring clothes (e.g., sports bra, halter top, or swimming suit, etc.) to expose the upper back/neck region, and will change into those in an isolated room and within the overall laboratory space. A gown will be provided for additional privacy.
5. Two researchers will be in the room during the session, with the gender of the researchers taken into account per participant. For example, for a male participant, the investigators plan to have a male researcher present during the session along with the female physical therapist. For a female participant, the investigators plan to have both the female physical therapist and a female researcher present.
6. The study team will apply non-toxic, washable ink to the participant's back in two 10 by 10 cm areas near the shoulder blades on either side of the body.
7. The participant will lie flat on a massage table.
8. A camera system will record the movements of the fingers of the physical therapist, along with the movements of the skin. The investigators will videotape the upper part of the participant's back. A participant's face will never be videotaped, nor will audio be recorded.
9. The physical therapist will conduct standard assessment procedures for about 2 minutes per side of the body, where the skin tissue will be compressed and slightly stretched
10. A soft tissue intervention, or massage, lasting about 15 minutes will take place in the participant's upper back/neck region.
11. Another assessment like that prior will be performed.
12. The participant will again be verbally asked about the current level of pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or diagnosed with benign, non-vascular headache and associated cervical musculoskeletal dysfunction (e.g. tender spots, trigger points, stiffness.
* Adult male and female.

Exclusion Criteria:

* Migraine headaches.
* Known cardiovascular, pulmonary, or metabolic disease.
* Any co-morbidities that could contribute to back or neck pain (e.g., head trauma, cancer, seizures, tumors, radiculopathies, rheumatoid arthritis, systemic auto-immune or inflammatory conditions).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Gerling, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in the area of soft tissue manipulation.
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact gg7h@virginia.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in January 2024 from university academic setting.
Pre-assignment Details: No pre-assignment exclusions were applied. All participants who enrolled proceeded directly to study assignment.
Groups:
- Manual Therapy Intervention: All participants with myofascial pain in the cervicothoracic region were assessed by a trained and licensed clinician, then received a standardized 15-minute manual therapy intervention. Outcomes were measured both immediately before and after the intervention to evaluate changes in tissue mobility and pain.
Period: Overall Study
Arm/Group | Manual Therapy Intervention
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Manual Therapy Intervention
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Self-reported pain [Mean (Standard Deviation); unit: Scores on a scale] — Pain self-reported on a scale of 0 (no pain) to 10 (worst pain) for cervicothoracic region.
  Scores on a scale | 3.4 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Skin Stretch Response to Manual Lateral Pull
Description: In the study overall, a non-invasive surface skin imaging technique with three cameras is used to determine soft tissue deformation and mobility. Using this basis of data, this outcome measure characterizes the skin's stretch response to the manual application of lateral pull perpendicular to it's surface, as the clinician pulls the tissue lateral to its surface with her fingertips. Therefore, from this data, the specific outcome measure is 1st principal strain (%) against manual pull (which is measured as maximum displacement, in units millimeters) for each of the two directions of pull (superior - towards neck, inferior - away from neck).
Time Frame: Measured once at start and once at finish of one hour session per participant
Measure: Mean (Standard Deviation); unit: %/mm
Arm/Group | Manual Therapy Intervention
Number analyzed (Participants) | 5
%/mm
  Superior direction, pre-intervention | 0.512 (0.131)
  Inferior direction, pre-intervention | 0.494 (0.128)
  Superior direction, post-intervention | 0.508 (0.178)
  Inferior direction, post-intervention | 0.473 (0.095)

2. Secondary Outcome: Clinical Evaluation of Range of Motion
Description: The assessing clinician will record the range of motion (ROM) of the neck with the subject in the upright, seated position, using a head mounted inclinometer system (Cervical Range-of-Motion Instrument Basic). Cervical ROM will be assessed bilaterally in four directions, a) extension, b) flexion, c) rotation, and d) lateral flexion. Units of degrees will be recorded per each motion.
Time Frame: Measured once at start and once at finish of one hour session per participant
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Manual Therapy Intervention
Number analyzed (Participants) | 5
Degrees
  Extension, pre-intervention | 62.40 (18.24)
  Flexion, pre-intervention | 43.60 (8.76)
  Rotation, pre-intervention | 54.70 (20.17)
  Lateral flexion, pre-intervention | 33.20 (9.81)
  Extension, post-intervention | 68.80 (16.77)
  Flexion, post-intervention | 47.20 (9.44)
  Rotation, post-intervention | 54.20 (18.91)
  Lateral flexion, post-intervention | 39.60 (12.64)

3. Secondary Outcome: Clinical Evaluation of Pressure Pain Threshold
Description: The assessing clinician will use Algometry to quantify pressure pain threshold (PPT), defined as the minimum pressure applied with a handheld algometer at which the sensation changed from pressure to discomfort. Units of Newtons will be recorded.
Time Frame: Measured once at start and once at finish of one hour session per participant
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Manual Therapy Intervention
Number analyzed (Participants) | 5
Newtons
  Pre-intervention | 32.10 (14.94)
  Post-intervention | 38.70 (14.31)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 1 week.
Description: Adverse events were monitored throughout the intervention and post-assessment period. The licensed clinician completed standardized post-intervention assessment and follow-up check-in with participants a few hours after treatment.
Arm/Group | Manual Therapy Intervention
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT06390085/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT06390085/SAP_001.pdf
  • Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT06390085/ICF_002.pdf